CLINICAL TRIAL: NCT00516230
Title: Establishing Effective Screening Methods for Diagnosing Hereditary Nonpolypoisis Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Other Study IDs: SMC-2007-04-080
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2007-08-15 (Estimated); Status verified 2007-08

CONDITIONS: Colonic Neoplasms
Keywords: Colonic Neoplasms; Lynch syndrome
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Correct identification of Lynch syndrome at the time of colorectal cancer presentation is important. We aim to find best ways to screen patients with colorectal cancer in Korea.

DETAILED DESCRIPTION:
Patients with newly diagnoised colorectal cancer will be eligible. They will undergo detailed history taking including family history, and molecular stuidies including microsatellite instability test and immunohistochemistry for DNA mismatch repair protein with pre-selection. Any abnormal finding in molecular stuides will be offered genetic testing (after testing methylation status for patients with abnormalities in MLH1).

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer

Exclusion Criteria:

* Histology showing other than adenocarcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-01; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Kyung Chang, M.D. Ph.D, Principal Investigator — Division of Gastroenterology, Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea